CLINICAL TRIAL: NCT06058104
Title: Evaluating Efficacy of a Digital Game Based Therapeutic for Improving Socialization Outcomes in Autistic Children, A Randomized Clinical Trial.
Brief Title: Evaluating Efficacy of a Digital Game Therapeutic for Children With Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dennis Paul Wall, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 60181-Stanford
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: digital; mobile health; autism; pediatrics
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: We will use block randomization stratified by sex to assign participants to the group where they will use the treatment immediately for 8 weeks or the cross over waitlist control, where they will be able to use the treatment after 8 weeks.
Who Masked: Investigator
Masking Description: The parent will know whether their child is receiving the treatment or not as they administer the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charades-based mobile digital therapeutic (Experimental): The mobile app is a charades style game and app that engages parent and child in fluid social interaction where the parent must guess what the child is acting out based on the prompt shown on the phone screen. Participants will use their own personal phone to download the study app. Parents are asked to play with their child for 15 minutes 3-4 times per week for 8 weeks.
  Interventions: Device: Charades based mobile digital therapeutic
- Treatment as Usual (No Intervention): Participants in control group will continue their Applied Behavior Analysis therapy as usual for 8 weeks, and then will be able to cross-over to the treatment condition at week 8.

INTERVENTIONS:
Device: Charades based mobile digital therapeutic — The mobile app is a charades style game and app that engages parent and child in fluid social interaction where the parent must guess what the child is acting out based on the prompt shown on the phone screen. Participants will use their own personal phone to download the study app. Parents are asked to play with their child 15 minutes 3-4 times per week for 8 weeks.
  Other Names: GuessWhat
  Arms: Charades-based mobile digital therapeutic

SUMMARY:
The following study aims to assess the efficacy of the game-based digital therapeutic, GuessWhat, in improving adaptive socialization skills in children with Autism Spectrum Disorder (ASD). GuessWhat is a mobile application (available for free for iOS and Android) which contains a suite of games: pro-social charades, emotion guessing, and quiz. Participant families will use their personal smartphones to download the app and play it with their child according to a predetermined regimen.

DETAILED DESCRIPTION:
The following study aims to understand the efficacy of the digital therapeutic, GuessWhat, in improving socialization outcomes in children with Autism Spectrum Disorder (ASD) after regular use over 8 weeks. We will use a cross-over, waitlist control design to examine outcomes after 8 weeks. GuessWhat is a mobile application (available for free for iOS and Android) which contains a suite of games: pro-social charades, emotion guessing, and quiz. Participant families will use their personal smartphones to download the app and play it with their child according to a predetermined regimen. The study will enroll parents who are at least 18 years old and have a child between 3 and 12 years old with a formal ASD diagnosis. Parents will be asked to complete two clinical outcome measure questionnaires immediately prior to and up to 1 week after playing GuessWhat with their child 3 times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Parent who is at least 18 years old of child with autism.
2. Child with autism is between 3 and 12 years old at time of baseline data collection.
3. A professional diagnosis of Autism that is able to be confirmed by negative score on a machine learning based algorithm using items from Mobile Autism Risk Assessment and video based classifier or by a copy of diagnostic report.

Exclusion Criteria:

1. Parent is unable to read the app in the offered languages (English, Spanish, Portuguese)
2. Parent does not have an Android or iOS smartphone compatible with GuessWhat App.
3. Child has additional psychiatric or neurologic diagnoses including genetic syndromes or epilepsy in addition to autism.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in parent reported socialization based on the Vineland Adaptive Behavior Scales 3rd Edition (VABS-3) Parent/Caregiver Socialization Subscale, from baseline to week 8 | Baseline (Week 0), Week 8
  Vineland Adaptive Behavior Scales, 3rd edition (VABS-3) Socialization subscale of the Parent/Caregiver Comprehensive form will be administered online to the parents. Scores from the socialization domain of the VABS-III reflects one's functioning in social situations. The socialization subscale is up to 112 items depending on age and development, where raw scores are converted to Intellectual Quotient-type standard scores--v-scale scores (M=15, SD=3) where scores range from 1 to 24, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning.

SECONDARY OUTCOMES:
Change in Parental Stress Scale - from baseline to week 8 | Baseline (Week 0), Week 8
  The Parental Stress Scale is an 18-item parent report scale that evaluates the extent of parent stress. Scores range from 18-90, where higher scores indicate a higher level of Parental stress.
Change in Emotion Recognition from baseline to week 8 | Baseline (Week 0), Week 8
  Study team will use an image based emotion recognition task where participants will select the emotion that corresponds to an emotional facial image in the form of a GIF (Graphics Interchange Format) image. Participants will select 1 of 8 available Ekman emotion labels for 16 facial emotional image stimuli presented in random order. Correct responses will be measured against a predetermined majority rules consensus of the emotional content of the GIFs.

OTHER OUTCOMES:
mobile autism risk assessment score at baseline | baseline (week 0)
  Study team will use a level 2 screening tool that has been validated in several studies and that uses a brief parent/caregiver questionnaire with a 2 minute home video to generate a classification score that indicates severity of the autism phenotype (ranging from no autistic symptoms to severe autism) as well as confidence in the classification.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Wall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT06058104/Prot_SAP_000.pdf